CLINICAL TRIAL: NCT06689826
Title: Investigation of the Relationship Between Core Muscle Strength, Balance and Dyskinesia in Patients With Unilateral Rotator Cuff Injury: Case Control Study
Brief Title: Investigation of Core Muscle Strength in Patients With Unilateral Rotator Cuff Injury
Status: Enrolling by invitation | Type: Observational
Sponsor: Ahi Evran University Education and Research Hospital (Other)
Responsible Party: Principal Investigator, Esra BAYRAMOĞLU DEMİRDÖĞEN, LECTURER DOCTOR, Ahi Evran University Education and Research Hospital
Other Study IDs: KAEU-EBAYRAMOGLUD-001; ESRA BAYRAMOĞLU DEMİRDÖĞEN (Registry Identifier: ESRA BD)
Record Dates: First submitted 2024-10-22; First posted 2024-11-14 (Actual); Last update posted 2024-11-20 (Actual); Status verified 2024-11

CONDITIONS: Shoulder Pain Chronic; Core Strength
Keywords: SHOULDER PAIN; CORE
MeSH Terms: conditions — Shoulder Pain

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Patient Registry: Yes
Target Follow-Up Duration: 1 Day
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- patient: Individuals diagnosed with unilateral rotator cuff

SUMMARY:
Located in the middle of the kinetic chain system, the core muscles are the regions where forces are generated and transferred to the extremities of the body. The core includes the abdominal muscles in the front, the paraspinal and gluteal muscles in the back, the diaphragm muscle above, and the pelvic floor and hip girdle muscles below. Good core function is essential for performing dynamic upper and lower extremity movements.

A relationship between shoulder function and the core region has been shown through the activation of core muscles during upper extremity movements. Muscle strength and endurance in the core region are needed to maintain functional stability during glenohumeral movements.

The ability to maintain shoulder function is largely dependent on the stability of the trunk, which is closely related to the stability and balance control of the lower extremities. The shoulder girdle needs to compensate for the loss of core stability and/or inadequate coordination of the legs, trunk, or scapula by increasing the speed and/or power of movement. There are studies showing that weight shifts to the affected side in patients with shoulder pain. However, it is not clear whether balance disorders in patients with shoulder pathology contribute to shoulder pathology or, more accurately, whether they are a result of shoulder pathology.

Changes in the static position of the scapula or dynamic scapular movement are generally defined as scapular dyskinesia. Due to changes in normal scapular kinematics, the normal biomechanics of the shoulder and joint stability also change. Scapular dyskinesia mostly occurs as a result of changes in coordination or activation between muscles.

As a result, investigators planned their study based on the fact that shoulder pathologies can affect core, balance and scapular dyskinesia. For this purpose, investigators will compare the measurements investigators will take from those with unilateral shoulder pain and healthy individuals.

DETAILED DESCRIPTION:
Grip Strength: Camry brand Digital Hand Dynamometer will be used for measurement. The measurement of hand grip strength will be made in the standard position recommended by the American Hand Therapists Association AETD; sitting position, shoulder adduction and neutral rotation, elbow 90 degrees flexion, forearm mid-rotation and support, wrist in neutral. According to the test procedure, 3 consecutive measurements will be made for hand grip strength and the averages will be recorded in kg. Pain: Visual Analog Scale will be used for pain assessment. This scale consists of a 10 cm horizontally positioned line on the page. The starting point on this line, '0', represents the patient feeling no pain, while the number '10' represents unbearable pain. The patient is asked to mark any place they want on this straight line between 0 and 10 to show the pain they have during the test. Then, the distance from the point marked by the patient to the starting point, 0, is measured with the help of a ruler and the value obtained is recorded. It will be questioned separately for rest and movement.

Core Strength: Measurements were made in 3 different positions with McGill Core Endurance Tests.

1. Trunk Flexion Test: The participant is asked to cross their hands on their chest. They are positioned on the floor with their body at 60° flexion and their knees at 90° flexion. The stopwatch is started. If there is any deterioration in their position, the stopwatch is stopped and the test is terminated. The elapsed time is recorded in seconds.
2. Side Bridge Test: The participant is asked to lie on their right side and place their foot on top of their other foot. They are asked to cross their left arm over their chest and place it on their right shoulder and rest on their right forearm and elbow. The stopwatch is started. If there is any deterioration in their position, the stopwatch is stopped and the test is terminated. The elapsed time is recorded in seconds. The same measurement is repeated for the left side.
3. Trunk Extensor Test: Participants are positioned in a prone position with their anterior superior iliac spines at the edge of the bed. Participants are asked to extend their upper bodies straight forward from the edge of the table. They are fixed on their knees with a belt. The stopwatch is started. If there is any deterioration in the position, the stopwatch is stopped and the test is terminated. The elapsed time is recorded in seconds.

Balance: Balance assessment will be performed with the Biodex Balance System (Biodex Medical Systems Inc., Shirley, New York, USA). The patient will be positioned on a platform with a screen in front of them. In our study, a rigid platform will be used and the patient will be given the appropriate position by holding on to the side bars with their hands while both feet (bare) are on the platform. The foot coordinates are determined while the patient is in the most comfortable position where they can maintain their balance. For the static postural balance measurement, patients are asked to hold the circular ring they see on the screen in the center for 20 seconds. The test is terminated after 3 measurements, each with 10 seconds of rest. Patients will repeat this measurement with their eyes open and closed.

Functionality: Functionality will be assessed with the Shoulder Pain and Disability Index (SPADI), which was developed for use in patients with shoulder pain and has been validated and reliable. Different activities are also used to assess pain and disability. It consists of 2 sections, pain and disability, and 13 questions. There are 5 questions in the pain section and 8 questions in the disability section. The score varies between 0 and 130. A high score indicates a high level of pain and disability.

Dyskinesia: Scapular dyskinesia will be assessed with the Lateral Scapular Slide Test.

Lateral Scapular Slide Test: Scapular position is measured by taking the side-to-side differences between both sides in all 3 test positions. Measurements are taken from the lower corner of the scapula to the spinous process of the thoracic vertebrae in the same horizontal plane.

The test is performed in 3 positions; Position 1: involves bringing the shoulders to a neutral position and relaxing the arms at the sides.

Position 2: The patient's hands are positioned around the waist and the humerus is placed in medial rotation and 45 degrees of abduction.

Position 3: The humerus is placed in maximum medial rotation and 90 degrees of abduction.

The test is positive when the measurements are compared bilaterally and there is a difference of 1.5 cm.

ELIGIBILITY:
Inclusion Criteria:

* Being between the ages of 18-65,
* Complaining of unilateral shoulder pain,
* Diagnosed with rotator cuff (Grade 1-2 rupture),
* Volunteer individuals who can cooperate

Exclusion Criteria:

* Presence of diabetes mellitus,
* Presence of a neurological problem,
* Presence of cervical disc herniation,
* Past history of orthopedic disease on the affected side,
* Presence of osteoarthritis, rheumatoid arthritis or any systemic inflammatory problem,

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: LIVING IN KIRSEHIR PROVINCE
Sampling Method: Probability Sample
Enrollment: 132 (Estimated)
Dates: Start 2024-08-16 (Actual); Primary Completion 2024-12-15 (Estimated); Study Completion 2024-12-25 (Estimated)

PRIMARY OUTCOMES:
core muscle strength | during the intervention.
  McGill Endurance Tests and Prone Bridge Test

SECONDARY OUTCOMES:
balance | during the intervention.
  Balance assessment will be performed with the Biodex Balance System (Biodex Medical Systems Inc., Shirley, New York, USA). The patient will be positioned on a platform with a screen in front of them. In our study, a rigid platform will be used and the patient will be positioned appropriately by holding onto the side bars with their hands while both feet (bare) are on the platform. The foot coordinates are determined while the patient is in the most comfortable position where they can maintain their balance. For static postural balance measurement, patients are asked to hold the circular ring they see on the screen in the center for 20 seconds. The test is terminated after 3 measurements including 10-second rest periods. Patients will repeat this measurement with their eyes open and closed.
grip strength | during the intervention.
  measurement of upper extremity muscle strength
Deviation of the scapula | during the intervention.
  It is a change or deviation from the normal, resting or active position of the scapula during shoulder movement.
Shoulder Pain and Disability Index (SPADI) | during the intervention.
  surveys

CONTACTS AND LOCATIONS:
Overall Officials: ESRA BAYRAMOGLU DEMIRDOGEN, LECTURER, Principal Investigator — Physiotherapist
Locations (1):
- Kirşehir Ahi Evran University Physical Therapy and Rehabilitation Hospital, Kırşehir, Centre, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
contains patient-specific data